CLINICAL TRIAL: NCT06212284
Title: General and Anxiety-Linked Influence of Acute Serotonin Reuptake Inhibition on Neural Responses Associated With Attended Visceral Sensation
Brief Title: Serotonin, Anxiety and Visceral Sensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sussex (Other)
Responsible Party: Principal Investigator, Daniel Campbell-Meiklejohn, Senior Lecturer, University of Sussex
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ER/JL332/9
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: serotonin; interoception; ssri; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- citalopram first, placebo second (Other): Citalopram was taken first. Placebo was taken at least 7 days later.
  Interventions: Drug: Citalopram 20mg; Drug: Placebo
- placebo first, citalopram second (Other): Placebo was taken first. Citalopram was taken at least 7 days later.
  Interventions: Drug: Citalopram 20mg; Drug: Placebo

INTERVENTIONS:
Drug: Citalopram 20mg — Doses were delivered in gelatine capsules filled with microcrystalline cellulose.
Drug: Placebo — Doses were gelatine capsules filled with microcrystalline cellulose

SUMMARY:
The goal of this crossover study was to learn about the potential regulatory role of serotonin in interoceptive processing and its relationship to levels of state anxiety. This experiment directly compared the impact of a selective serotonin reuptake inhibitor (SSRI) (20mg CITALOPRAM) to that of a PLACEBO on the neural processing of ordinary interoceptive sensations and the relationship of these influences to anxious states.

Healthy young volunteers completed the visceral interoceptive attention task with each treatment condition (citalopram and placebo). The task involves focusing attention on heart, stomach, or visual sensation control while scanned with functional magnetic resonance imaging (fMRI). The difference in haemodynamic response between interoceptive sensation(s) and visual sensation (i.e. the relative interoceptive response) is compared between treatment conditions. State anxiety is measured at each test period. It is used to test for a moderating effect of state anxiety on the influence of serotonin in interoceptive processing and used post-hoc to explore associations between changes in state anxiety and changes of interoceptive relative interoceptive response due to the SSRI.

ELIGIBILITY:
Inclusion Criteria:

- healthy volunteer

Exclusion criteria included:

* the presence of significant ongoing medical condition;
* pregnancy or breastfeeding;
* currently taking any medication (excluding contraceptive pill);
* first-degree family history of bipolar disorder;
* an indication of current or historical mental health disorder,
* MRI scanner contraindications (e.g. metallic implants)
* data that is unanalyzable due to movement
* excessive side effects of the drug (e.g. nausea)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-02-18 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
relative neural interoceptive response - heart | 15 minutes
  Neural response, inferred via functional magnetic resonance imaging from focusing attention on the heart, minus the response during focus on a visual stimulus
relative neural interoceptive response - stomach | 15 minutes
  Neural response, inferred via functional magnetic resonance imaging from focusing attention on the stomach, minus the response during focus on a visual stimulus
State Anxiety | 5 minutes
  State Trait Anxiety Inventory

SECONDARY OUTCOMES:
Metacognitive Interoceptive Insight | 45 minutes
  Ability of confidence to predict accuracy when making decisions about whether heartbeat is in sync with an auditory tone. This is an exploratory measure.
Physiological and Psychological state | Measured twice, for 2 minutes, before and after scanning. Average taken to estimate state inside scanner.
  Three scales (from 0-100) were given to assess three somatic side effects (nausea, headache and dizziness). Five anxiety-related effects (pairs of antonyms: alert-drowsy, stimulated-sedated, restless-peaceful, irritable-good-humoured, anxious-calm) were used to confirm other anxiety measures and alert the researchers to excessive side effects. Used to confirm anxiety measure detect side effects.
Positive and Negative Affect Scale | Measured twice, for 2 minutes, before and after scanning. Average taken to estimate state inside scanner.
  Measures affective state, confirming anxiety measure
Heartrate | Before scans of each session, 2 minutes
  Participants had their heartrate recorded with the participant relaxed and sitting.
Cerebral Blood Flow Change | 2 minutes, at scan
  Perfusion imaging, to control for effects of citalopram on blood flow
Anatomical scan and fieldmaps | 6 minutes, at scan
  For coregistration of functional magnetic resonance images

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Campbell-Meiklejohn, DPhil, Principal Investigator — University of Sussex
Locations (1):
- School of Psychology, Falmer, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared on a publically accessible database with a link accessible through the official publication.
Time Frame: After publication
Access Criteria: Public Access